CLINICAL TRIAL: NCT07230548
Title: Effect of Single Instillation of Four Different Diagnostic Eye Drops on Tear Film Thickness in Healthy Subjects
Brief Title: Effect of Four Different Diagnostic Eye Drops on Tear Film Thickness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Doreen Schmidl, Assoc.Prof. PD Dr., PhD, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: OPHT-250618
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Ocular Surface Disease; Tear Film Characteristics
MeSH Terms: interventions — benoxinate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oxybuprocaine MDU (Active Comparator): Subjects will receive 30µl of oxybuprocaine preserved in multi-dose units (MDU) in both eyes after the baseline measurements on the randomized study day
  Interventions: Drug: Oxybuprocaine MDU
- Oxybuprocaine SDU (Active Comparator): Subjects will receive 30µl of oxybuprocaine preserved in single-dose units (SDU) in both eyes after the baseline measurements on the randomized study day
  Interventions: Drug: Oxybuprocaine SDU
- Fluorescein SDU (Active Comparator): Subjects will receive 30µl of fluorescein preserved in single-dose units (SDU) in both eyes after the baseline measurements on the randomized study day
  Interventions: Drug: Fluorescein SDU
- Oxybuprocaine/fluorescein SDU (Active Comparator): Subjects will receive 30µl of oxybuprocaine/fluorescein preserved in single-dose units (SDU) in both eyes after the baseline measurements on the randomized study day
  Interventions: Drug: Oxybuprocaine/fluorescein SDU

INTERVENTIONS:
Drug: Oxybuprocaine MDU — the effect of instillation of 30µl of oxybuprocaine preserved as multi-dose unit (MDU) in both eyes will be investigated
  Arms: Oxybuprocaine MDU
Drug: Oxybuprocaine SDU — the effect of instillation of 30µl of oxybuprocaine preserved as single-dose unit (SDU) in both eyes will be investigated
  Arms: Oxybuprocaine SDU
Drug: Oxybuprocaine/fluorescein SDU — the effect of instillation of 30µl of oxybuprocaine/fluorescein preserved as single-dose unit (SDU) in both eyes will be investigated
  Arms: Oxybuprocaine/fluorescein SDU
Drug: Fluorescein SDU — the effect of instillation of 30µl of fluorescein preserved as single-dose unit (SDU) in both eyes will be investigated
  Arms: Fluorescein SDU

SUMMARY:
The use of topical anesthesia as well as corneal vital staining with fluorescein is an inevitable part of various ophthalmological examinations and surgical treatments. However, eye drops that don't come in single dose packages are required to contain preservatives such as chlorhexidine diacetate. An increasing number of surveys proves the partly severe side effects that preservative-containing eye drops may induce. The aim of the present study therefore is to investigate the effects of four different topical diagnostic eye drops (Novain®, Minims Oxybuprocaine Hydrochloride®, Thilorbin® and Minims®) on tear film thickness in healthy subjects. Tear film thickness will be measured at baseline and at defined time points after single instillation. The course of tear film thickness during the study day will provide information about the influence on tear film stability of the four different eye drops. Healthy subjects will receive Novain®, Minims Oxybuprocaine Hydrochloride®, Thilorbin® and Minims® eye drops on 4 different study days in a randomized order. Assessment of lipid layer thickness will be performed before and at pre-specified time points after instillation as secondary outcome. Other clinical measures such as determination of tear film break up time (TFBUT), corneal sensation, and Schirmer I test will be performed. The study will be conducted in a randomized, single masked, observer blinded four-way cross-over design. Subjects will receive all four diagnostic eye drops on 4 different study days in a randomized order.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged at least 18 years
* Written informed consent prior to study-related procedures
* Normal ophthalmic findings
* No use of eye drops including topical lubricants in the 4 weeks before screening

Exclusion Criteria:

* Participation in a clinical trial in the 3 weeks preceding the study
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Presence or history of a severe medical condition as judged by the clinical investigator
* Intake of parasympathomimetic or anti-psychotic drugs
* Wearing of contact lenses
* Dry eye syndrome (Schirmer I test ≤10mm or TFBUT <10 sec.)
* Glaucoma in the medical history
* Treatment with corticosteroids in the 4 weeks preceding the study
* Topical treatment with any ophthalmic drug in the 4 weeks preceding the study
* Ocular infection or clinically significant inflammation
* Ocular surgery in the 3 months preceding the study
* Sjögren's syndrome
* Stevens-Johnson syndrome
* History of allergic conjunctivitis
* Pregnancy, planned pregnancy or lactating
* Known hypersensitivity to any component of the study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Change of tear film thickness | Predose and at defined time points (10±5, 20±5, 40±5, 60±5, 120±10 and 240±10 minutes) after single instillation
  Change of tear film thickness as measured with optical coherence tomography predose and at defined time points (10±5, 20±5, 40±5, 60±5, 120±10 and 240±10 minutes) after single instillation

SECONDARY OUTCOMES:
Corneal Sensation | Predose and at defined time points (10±5, 20±5, 40±5, 60±5, 120±10 and 240±10 minutes) after single instillation
  The measurement of corneal sensation predose and at defined time points (10±5, 20±5, 40±5, 60±5, 120±10 and 240±10 minutes) after single instillation using a Cochet-Bonnet aesthesiometer
Tear film break up time | Change of tear film break up time predose 240±10 minutes after single instillation
  Change of tear film break up time from baseline to 240±10 minutes after single instillation
Schirmer 1 test | Baseline to 240±10 minutes after single instillation
  Change of Schirmer 1 test as measured from baseline to 240±10 minutes after single instillation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided
The data that support the findings of this study are available from the corresponding author upon reasonable request.